CLINICAL TRIAL: NCT02547246
Title: Transcranial Magnetic Stimulation, Embodied Cognition and Bulimic Craving
Brief Title: Transcranial Magnetic Stimulation and Bulimic Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1108053; 2011-A00481-40 (Other: ANSM)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Bulimia
Keywords: bulimia; repetitive transcranial magnetic stimulation (rTMS)
MeSH Terms: conditions — Bulimia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS session (Experimental): Patients will have a 20 minute session of rTMS at a frequency of 10 Hz.
  Interventions: Device: rTMS session
- rTMS placebo (SHAM) session (Placebo Comparator): Patients will have a 20 minute session of placebo rTMS
  Interventions: Device: rTMS Placebo (SHAM)

INTERVENTIONS:
Device: rTMS session — One session of rTMS at a frequency of 10 Hz during 20 minutes
  Arms: rTMS session
Device: rTMS Placebo (SHAM) — One session of placebo (SHAM) rTMS during 20 minutes
  Arms: rTMS placebo (SHAM) session

SUMMARY:
Bulimic patients suffering from binge eating or "craving" a pressing need to eat, with a sense of unease and anxiety, relieved by food intake. The phenomenon of craving bulimia may be considered appropriately by using paradigms developed in the framework of embodied cognition theories.

In bulimic, a study with 20 bulimic patients proved an automatic attraction (unconscious) for food in these patients, as measured by reaction time.

Moreover, a therapeutic explored in bulimia (particularly on reducing craving), is repeated transcranial magnetic stimulation (rTMS). Studies have shown that a single session of rTMS to the dorsolateral prefrontal cortex left (DLPFC) reduces significantly the food craving among bulimics, 24 hours after stimulation. But the therapeutic efficacy of TMS on bulimia to more than 24 hours has not yet been demonstrated, and the psycho-cognitive underlying mechanisms have not yet been explored.

DETAILED DESCRIPTION:
The exams / treatments of the study include:

* a 20 minute session of rTMS at a frequency of 10 Hz.
* cognitive testing and attention, which will be made on the computer before and 24 hours after the session of rTMS.

Cognitive test consist in , on a computer screen:

* Is first displayed, food and non-food words. The patient must pull a lever to it if the letter A is present in the word and push the lever if the letter A is missing the word.
* Then presents a series of food and non-food words. The patient must pull a lever to it if it deems that the word has a positive meaning and push the lever if it determines that the word has a negative meaning

ELIGIBILITY:
Inclusion Criteria:

* right-handed patient
* Patients without psychotropic treatment or treatment with a stable and unchanged for over a month.
* Normal BMI

Exclusion Criteria:

* Previous history of seizures or epilepsy.
* Participants with a somatic problem restricted movement or an uncorrected visual acuity problem.
* History of head trauma, neurological disease or unstabilized serious physical illness.
* Major Depressive Episode at the time of the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Motor response time | 24h after rTMS session
  time taken to pull or push the lever in cognitive tests (composite measure)

CONTACTS AND LOCATIONS:
Overall Officials: Torrance SIGAUD, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No